CLINICAL TRIAL: NCT02341976
Title: Study of Pelvic Floor Muscle and Urinary Sphincter Activity by Electromyography During Whole Body Vibration Training
Brief Title: Whole Body Vibration Training for Pelvic Floor Muscle
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left University and no study was ever done
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1405M50481
Record Dates: First submitted 2014-05-27; First posted 2015-01-19 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: whole body vibration; pelvic floor muscle; urinary incontinence; Urinary sphincter
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vibratory platform exercises (Other): Vibratory platform exercises: different positions on a vibratory platform in different frequencies
  Interventions: Other: Vibratory platform exercises

INTERVENTIONS:
Other: Vibratory platform exercises — Different positions on vibratory platform with different frequencies

SUMMARY:
To study which position on the whole body vibrator machine would stimulate the pelvic floor muscles.

DETAILED DESCRIPTION:
Urinary incontinence is a common problem due to a weak pelvic floor muscle associated with decrease quality of life. The vibration exercises have been associated with improvements of the muscle component. Due to this, some researches have proposed that this technique could be applied to weak pelvic floor. However, it is unknown which vibration trainings have the highest impact on the pelvic floor muscle and urinary sphincter, more objectives studies to validate these data are necessary.

The purpose of our research is to evaluate the activity in the urinary sphincter and the pelvic floor muscle by vibratory platform training in women.

Subjects will be recruited, criteria exclusion will be evaluated, age, and BMI will be recorded. Each subject will exercise on the vibratory platform in 3 different positions, each one with 2 different frequencies and 1 minute each position and frequency. Pelvic electromyography (EMG) will assess the activity of the urinary sphincter and pelvic floor muscle with vibratory exercise. Data will be collected during all procedures.

According to our purpose and anticipating the impact of this research extrapolating whole body vibration (WBV) training as program to improve the strength of the pelvic floor muscle elaborating a guided plan to improve clinical outcomes and quality of life of patients suffering from urinary incontinence with this new nonsurgical treatment approach to women with mild to moderate stress urinary incontinence, as well as this research allow us to increase our knowledge in urinary continence and the pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

Women over 18 years of age

Exclusion Criteria:

Criteria exclusion like unhealthy condition, acute thrombosis, acute inflammations, implants, fractures, acute tendinopathies, kidney or bladder stones, gallstones, lung disease, heart disease, skin disease, hypertension, any medication or disease known to affect muscle mass or strength and pregnant will be evaluated

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Peak average of the pelvic floor activity (measured by Electromyography (EMG) | 1 year
  The primary assessment that will be reported will evaluate the mean of the peak activity measured by Electromyography (EMG) reached by the different exercises

SECONDARY OUTCOMES:
Proportion of the Maximum Voluntary contraction (MVC) peak average reached by the peak average of the muscle contraction with each Whole Body Vibration (WBV) exercise | 1 year
  The second assessment that will also be reported will evaluate the proportion of the MVC peak average reached by the peak average of the muscle contraction with each WBV exercise. A positive impact of the exercise will be considered if this reaches over 60% of the MVC. On the other hand, the investigators will define as no impact when below 60% of the MVC is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Nissrine Nakib, MD, Principal Investigator — University of Minnesota

REFERENCES:
- [Result] Petros PE, Ulmsten UI. An integral theory and its method for the diagnosis and management of female urinary incontinence. Scand J Urol Nephrol Suppl. 1993;153:1-93. No abstract available. PMID 8108659
- [Result] Marin PJ, Ferrero CM, Menendez H, Martin J, Herrero AJ. Effects of whole-body vibration on muscle architecture, muscle strength, and balance in stroke patients: a randomized controlled trial. Am J Phys Med Rehabil. 2013 Oct;92(10):881-8. doi: 10.1097/PHM.0b013e318292336c. PMID 23636085
- [Result] Maikala RV, King S, Bhambhani YN. Acute physiological responses in healthy men during whole-body vibration. Int Arch Occup Environ Health. 2006 Feb;79(2):103-14. doi: 10.1007/s00420-005-0029-8. Epub 2005 Sep 21. PMID 16175416
- [Result] Mikhael M, Orr R, Fiatarone Singh MA. The effect of whole body vibration exposure on muscle or bone morphology and function in older adults: a systematic review of the literature. Maturitas. 2010 Jun;66(2):150-7. doi: 10.1016/j.maturitas.2010.01.013. Epub 2010 Feb 19. PMID 20171817
- [Result] Machado A, Garcia-Lopez D, Gonzalez-Gallego J, Garatachea N. Whole-body vibration training increases muscle strength and mass in older women: a randomized-controlled trial. Scand J Med Sci Sports. 2010 Apr;20(2):200-7. doi: 10.1111/j.1600-0838.2009.00919.x. Epub 2009 Apr 20. PMID 19422657